CLINICAL TRIAL: NCT04743050
Title: The Use of Alpha-linolenic (ALA), Docosahexaenoic (DHA) and Eicosapanthene (EPA) Esters in the Prevention of Cardiovascular Diseases in Adults.
Brief Title: The ALA, DHA and EPA Esters in the Prevention of Cardiovascular Diseases.
Acronym: OMEGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KB-596/2020
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-12

CONDITIONS: Fatty Acids; Alpha-Linolenic Acid; Docosahexaenoic Acids; Eicosapentaenoic Acid; Preventive Health Services; Preventive Medicine; Cardiovascular Diseases; Anti-Inflammatory Agents
Keywords: Essential polyunsaturated fatty acids; EFA; EFAs; ALA; EPA; DHA; Esters
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fatty Acids, Unsaturated; Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): The control group will be a group without EFA supplementation.
  Interventions: Diagnostic Test: Diagnostic Tests
- 1st Experimental Group (Experimental): The first experimental group will receive supplementation with pure ALA fraction of EFA esters. 5 ml a day of OmegaRegen Original containing 2.9 g of ALA, 0.9 g of oleic acid and 0.8 g of linoleic acid for six months.
  Interventions: Drug: Fatty Acids, Unsaturated; Diagnostic Test: Diagnostic Tests
- 2nd Experimental Group (Experimental): The second test group will receive supplementation of the EPA and DHA fraction of EFA esters. 5 ml a day of OmegaRegen EPA+DHA containing 0.032 g of EPA, 0.192 g of DHA, 0.9 g of oleic acid and 0.8 g of linoleic acid for six months.
  Interventions: Drug: Fatty Acids, Unsaturated; Diagnostic Test: Diagnostic Tests
- 3rd Experimental Group (Experimental): The second test group will receive supplementation of the EPA and DHA fraction of EFA esters. 5 ml a day of OmegaRegen MAMA containing 2.9 g of ALA, 0.032 g of EPA, 0.192 g of DHA, 0.9 g of oleic acid and 0.8 g of linoleic acid for six months.
  Interventions: Drug: Fatty Acids, Unsaturated; Diagnostic Test: Diagnostic Tests

INTERVENTIONS:
Drug: Fatty Acids, Unsaturated — All participants from Experimental Groups will receive supplementation of different fractions of EFAs esters for six months daily. Control Group will be monitored with the same tests, but will not receive any supplementation.
  Other Names: OmegaRegen; Esters of Unsaturated Fatty Acids; EFA
  Arms: 1st Experimental Group; 2nd Experimental Group; 3rd Experimental Group
Diagnostic Test: Diagnostic Tests — All participants will have laboratory tests marking: CRP, fasting glucose, lipid profile, total blood count, and additional tests, which will include blood pressure measurements and measurements of body mass and composition on a specialized body composition analyzer (InBody 270). All the mentioned tests will be performed at the time of joining the research program, after 3 months (in the middle of the research program) and after 6 months (at the end of the research program).
  Other Names: Laboratory and Additional Tests

SUMMARY:
Essential polyunsaturated fatty acids (EFAs) have a significant impact on human health, even before birth. Their supplementation is recommended at all ages, especially in people with cardiolovascular risks. The most valuable proven action of EFAs is the improvement of the lipid profile (including increase in HDL, the so-called "good cholesterol" and lowering LDL, the so-called "bad cholesterol"), preventing the development of atherosclerosis, strokes and heart attacks.

We distinguish three fractions of EFAs: EPA, DHA and ALA. The best known are EPA and DHA, but in recent years the interest in ALA fraction has increased, as it is the only fraction that has pronounced anti-inflammatory properties, but also only ALA is not produced by the human body and must be supplied with food.

We believe that the supplementation of the ALA fraction is as important as the supplementation of the well-known and recommended EPA and DHA fractions, moreover it also brings unique benefits. The aim of the study is to demonstrate the benefits of EFAs in the prevention of cardiovascular diseases in the group of adults. In the project, we also want to compare the benefits of supplementing various fractions.

Each volunteer will be randomly assigned to one of 4 groups. Group No. 1 will be a group without the supplementation of essential fatty acids (EFAs), group No. 2 will receive supplementation with pure ALA fraction, group No. 3 will receive supplementation with EPA and DHA fractions, and group No. 4 will receive supplementation with all fractions, i.e. ALA, EPA and DHA. All persons from groups 1-4 will be examined three times: at the beginning, after three months and after six months (at the end of the project). The tests will include: blood pressure measurements, non-invasive measurements of body mass and composition, and laboratory tests: CRP, fasting glucose, lipid profile, and blood count.

Both preparations for acid supplementation and tests are completely free for participants.

Participation in the study is voluntary and is not associated with any health risk.

DETAILED DESCRIPTION:
Supplementation of essential polyunsaturated fatty acids (EFAs) in patients is recommended by cardiological, diabetic, hypertensive and gynecological societies. The project aims to demonstrate the benefits of following these recommendations in the prevention of cardiovascular diseases in the adult group. Most of the research focuses only on EPA and DHA fractions, while in view of the publications on the health-promoting properties of the ALA fraction, which is the only one that is only exogenous and has clear anti-inflammatory properties, in the project we also want to compare the benefits of supplementation of esters of individual EFA fractions. We intend to conduct a clinical trial with a control sample and 3 study groups randomly assigned to each group. The groups will consist of 50 people, which means that the research project will involve 200 people in total. The control group will be a group without EFA supplementation, the first experimental group will receive supplementation with pure ALA fraction of EFAs esters, the second experimental group will receive supplementation of the EPA and DHA fraction of EFAs esters, and the third experimental group will receive supplementation of the ALA, EPA and DHA fraction of EFAs esters. All participants will have laboratory tests marking: CRP, fasting glucose, lipid profile, total blood count, and additional tests, which will include blood pressure measurements and measurements of body mass and composition on a specialized body composition analyzer (InBody 270). All the above-mentioned tests will be performed at the time of joining the research program, after 3 months (in the middle of the research program) and after 6 months (at the end of the research program).

The aim of the study is to determine whether the supplementation of the ALA fraction esters of essential polyunsaturated fatty acids is as important as the supplementation of their EPA and DHA fraction esters, and whether it brings additional unique benefits related to its pronounced anti-inflammatory properties. This comparison is particularly important in the group of adults, as early and effective intervention may contribute to improving health, quality of life, increasing life expectancy and reducing treatment costs, and cardiovascular diseases as lifestyle diseases are one of the most common in the world and concern younger and younger people. The project's feasibility is assessed positively as the project has significant scientific potential. The discussed topic is up-to-date and the size of the studied group guarantees reliable results and gathering such a group remains possible. The importance of using EFAs in medicine is constantly increasing, and research using them gives promising results.

ELIGIBILITY:
Inclusion Criteria:

* adults of both sexes in good general condition.

Exclusion Criteria:

* pregnancy, acute diseases or uncontrolled / unchecked chronic diseases, indications for absolute treatment with lipid-lowering drugs or its modification, insulin-dependent diabetes mellitus, liver diseases, use of warfarin or heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Better glucose tolerance. | 6 months
  Decrease/normalization in fasting glucose level.
Improvement in lipid metabolism. | 6 months
  Decrease/normalization in lipid profile.
Lowering inflammatory markers. | 6 months
  Decrease of inflammatory markers.
Lowering blood pressure. | 6 months
  Decrease/normalization of blood pressure.
Improving blood count parameters | 6 months
  Normalization of total blood count values.
Lowering body weight. | 6 months
  Decrease of body weight, especially visceral adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Bujnowska-Fedak, MD, PhD, Study Director — Departament of Family Medicine at Wroclaw Medical University
Locations (3):
- Poland (3):
  - Department of Family Medicine at Wroclaw Medical University, Wroclaw, Dolny Slask
  - Model Practice of a Family Doctor Maria Bujnowska-Fedak, Wroclaw, Dolny Slask
  - TIGmed Private Medical Practice, Wroclaw, Dolny Slask

IPD SHARING:
Plan to Share IPD: No